CLINICAL TRIAL: NCT07306884
Title: Neurophysiological, Autonomic, and Sonographic Assessment of Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Rageh Daifallah Galal, Resident at Neurology and Psychiatry Department, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 09-2025-200567
Record Dates: First submitted 2025-09-25; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Diabete Mellitus; Peripheral (Sensorimotor) Diabetic Polyneuropathy
Keywords: Diabete Mellitus; Peripheral neuropathy; Neurophysiological studies; Nerve ultrasound; automatic assessment
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies; Peripheral Nervous System Diseases | interventions — Nerve Conduction Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetic patients with symptomatic peripheral neuropathy. (Other)
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Nerve ultrasound
- Diabetic without any clinical features nor complaints of peripheral neuropathy (Other)
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Nerve ultrasound; Diagnostic Test: Autonomic assessment
- Healthy individuals. (Other)
  Interventions: Diagnostic Test: Nerve conduction study; Diagnostic Test: Nerve ultrasound; Diagnostic Test: Autonomic assessment

INTERVENTIONS:
Diagnostic Test: Nerve conduction study — Nerve conduction studies (NCS) are widely regarded as the gold standard for evaluating large-fiber peripheral nerve function. They measure conduction velocity, latency, and amplitude, providing objective evidence of axonal loss or demyelination. While highly specific, NCS often detect abnormalities only in established diabetic peripheral neuropathy, limiting their sensitivity for early or subclinical disease.
Diagnostic Test: Nerve ultrasound — High-resolution ultrasound (HRUS) is a non-invasive imaging tool that allows structural evaluation of peripheral nerves. It can measure cross-sectional area (CSA), visualize fascicular pattern, and detect nerve enlargement or structural abnormalities. In diabetic peripheral neuropathy, HRUS provides complementary information to functional tests and may identify early or subclinical changes.
Diagnostic Test: Autonomic assessment — Autonomic testing provides insight into small-fiber and autonomic nervous system function, often impaired early in diabetic peripheral neuropathy. Heart rate variability (HRV) during deep breathing and postural change is a simple, non-invasive method to detect cardiovascular autonomic dysfunction
  Arms: Diabetic without any clinical features nor complaints of peripheral neuropathy; Healthy individuals.

SUMMARY:
Diabetic peripheral neuropathy causes pain, sensory loss, and foot risk; multimodal assessment enables earlier diagnosis and improved patient management.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) is a prevalent and disabling complication of diabetes, associated with pain, sensory deficits, gait instability, and increased risk of foot ulcers and amputation. Conventional diagnostic methods, such as nerve conduction studies, primarily identify established disease and may overlook early or autonomic involvement. A multimodal assessment integrating neurophysiological, autonomic, and sonographic techniques offers the potential for earlier detection, improved diagnostic accuracy, and optimized patient management.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-75 years with type 1 or type 2 diabetes (with or without diabetic peripheral neuropathy), and age and sex-matched healthy controls

Exclusion Criteria:

* Other causes of neuropathy (e.g., CIDP, trauma, toxins, vitamin deficiencies), advanced renal failure,thyroid disease,chronic alcohol use, pregnancy,
* presence of implanted cardiac devicesthat may interfere with autonomic testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of nerve conduction studies for diagnosing diabetic peripheral neuropathy | Baseline (single study visit)
  Percentage of participants with clinically diagnosed diabetic peripheral neuropathy who have abnormal nerve conduction study results (reduced amplitude and/or reduced conduction velocity) at the baseline visit.

SECONDARY OUTCOMES:
Correlation between tibial nerve cross-sectional area and tibial motor conduction velocity | Baseline (single study visit)
  Correlation coefficient between tibial nerve cross-sectional area measured by high-resolution ultrasound and tibial motor nerve conduction velocity at the baseline visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nageh Fouly, Study Chair — Department of Neurology , Assiut University, Egypt
Locations (1):
- Department of Neurology, Faculty of Medicine,Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided